CLINICAL TRIAL: NCT06849271
Title: HYbrid RObotic Surgery MulTiCentric Study (HYROS-MTC-I)
Brief Title: HYbrid RObotic Surgery MulTiCentric Study
Acronym: HYROS-MTC-I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rob Surgical Systems S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PL-PR01-150
Record Dates: First submitted 2025-01-09; First posted 2025-02-27 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Nephrectomy; Prostatectomy
Keywords: Radical nephrectomy; Partial nephrectomy; Radical prostatectomy; Lymphadenectomy; Lysis of adhesions; Robotic surgery; Minimal Invasive surgery; Minimal Invasive robotic surgery; Urology

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients surgically treated with ROB-Bitrack System and ESE/ NESE instruments and accessories (Experimental)
  Interventions: Procedure: Radical Nephrectomy (RN); Procedure: Partial nephrectomy (PN); Procedure: Radical Prostatectomy (RP)

INTERVENTIONS:
Procedure: Radical Nephrectomy (RN) — Complete remove of the kidney. In addition as part of the intervention, a procedure termed "Lysis of abdominal adhesions" may be performed according to patient medical condition and/or surgeon criteria.
Procedure: Partial nephrectomy (PN) — Partial remove of a section in the kidney. In addition, as part of the intervention, a procedure termed "Lysis of abdominal adhesions" may be performed according to patient medical condition and/or surgeon criteria.
Procedure: Radical Prostatectomy (RP) — Complete remove of the prostate gland. In addition as part of the intervention, two procedures termed "Lysis of abdominal adhesions" and/or "Lymphadenectomy " (removal of regional lymph nodes) may be performed according to patient medical condition and/or surgeon criteria.

SUMMARY:
The purpose of this clinical investigation, HYROS-MTC-I, is to confirm the effectiveness of the combined use of ROB-Bitrack System, its corresponding ElectroSurgical Endoscopic instruments and Non-ElectroSurgical Endoscopic instruments (ESE and NESE instruments respectively) and accessories in a multicentric study in urologic procedures with the indication of a robot assisted laparoscopic Radical/simple nephrectomy (RN), Partial nephrectomy (PN), Radical Prostatectomy (RP or P), and when it applies Lysis of Adhesions (during a PN, RN or RP or P to cut the adhesions and reach the organ) and Lymphadenectomy (only after a P with the aim to remove the lymph nodes) . HYROS-MTC-I is a confirmatory study in which the hypothesis of the primary endpoint is that: "Operative time (OT) with Bitrack System and its ESE/NESE Instruments and accessories will be equal or lower than superiority margin time of State of the Art (SoTA) of MIRS (Minimally Invasive Robotic Surgery) independently of the user experience and site". This study includes the data collected up to 30 days post-surgery.

DETAILED DESCRIPTION:
The ROB-Bitrack System is 4-arms on demand open and portable robotic platform indicated to be used during general abdominal laparoscopic surgical procedures. This robot is intended to assist in the accurate control of endoscopic instruments and accessories for endoscopic visualization and manipulation of tissue. The HYROS-MTC-I clinical investigation will be conducted as a multi-center, with a single arm, open-label, and non-randomized design, that will include 50 patients. The study shall refer to effectiveness of ROB-Bitrack System together with its accessories and corresponding ESE/NESE instruments. The planned visits for this clinical investigation are baseline (includes Screening, baseline visit, and Informed consent), procedure, discharge, 14-Days and 30-Days Follow-up visit . The clinical investigation will include adult subjects (between 18 and 90 years old) who have been scheduled for laparoscopic Radical Nephrectomy, Partial Nephrectomy or Radical Prostatectomy. The expected duration of the study is 12 months from the first patient enrolled, including 11 months of enrollment and the follow up of 30 days after surgery. The end of the clinical investigation will occur when the last visit of the last enrolled subject is completed.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects between 18 and 90 years old who have provided written informed consent prior to any clinical investigation related procedures.
2. Subjects who have been scheduled for a laparoscopic Radical/simple Nephrectomy surgery, laparoscopic Partial Nephrectomy or laparoscopic Radical Prostatectomy following the surgeon criteria.
3. Ability and willingness to comply with all study requirements to be evaluated for each study visit.

Exclusion Criteria:

1. Pregnant or breastfeeding women at the time of the surgery.
2. Subjects with severe concomitant illness that, at PrincipaI investigator´s discretion, increases risk of therapeutic interventions or that have been submitted to multiple prior surgeries.
3. Subjects admitted to the hospital due to an emergency situation.
4. Subjects with untreated active infection.
5. Subject with known allergy to some of the device components (i.e., stainless steel, etc.)
6. Subjects not suitable to undergo Minimally Invasive Surgery (MIS)/ Minimally Invasive Robotic Surgery (MIRS), according to medical criteria.
7. Subjects with life expectancy inferior to 3 months.
8. Subjects with a BMI (Body Mass Index) ≥ 40
9. Subjects with any contraindication for the use of the ROB-Bitrack System and the ESE/NESE instruments, as specified in the Instructions For Use.
10. Subjects with abuses of active substances or with uncontrolled psychiatric disorders.
11. Subjects with severe cardiopulmonary or coronary artery disease, bleeding disorders or that have been submitted to multiple prior operations.
12. Subjects scheduled for surgeries intended to be in direct contact with the heart, the central circulatory system or the central nervous system.
13. Inability to adhere to study-related procedures.
14. Subjects who participate in another trial which may affect the outcome data on this study or the ability to complete the follow up requirements

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Operative time (OT) with ROB-Bitrack System and its ESE/NESE Instruments and accessories to perform the surgeries. | During the procedure
  Evaluation of Operative time from first skin incision to last skin suture of the procedure.It is hypothesized that Operative time (OT) will be equal or lower than the maximum time as defined by the State of the Art (SoTA) of MIRS independently of the user experience and site.

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital del Mar, Barcelona, Spain
  - Hospital Clinic de Barcelona, Barcelona, Spain
  - Hospital General de Granollers, Granollers, Spain
  - Hospital de Mataró, Mataró, Spain
  - Hospital Universitari de Vic, Vic, Spain